CLINICAL TRIAL: NCT04978818
Title: Immunogenicity of H. Influenzae Type b PRP-OMP Vaccines in American Indian and Alaska Native Children
Brief Title: Immunogenicity of H. Influenzae Type b PRP-OMP Vaccines in American Indian and Alaska Native Children (the HibVax Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00011170
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Haemophilus Influenzae Type B Infection
Keywords: Native American; Vaccine
MeSH Terms: conditions — Haemophilus Infections | interventions — Vaxelis; Methods; Haemophilus influenzae-type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine

STUDY DESIGN:
Intervention Model Description: Randomization of participants will be done at the site level. Participants will be assigned randomly 1:1, to the Vaxelis arm or the PedvaxHIB arm. This is an unblinded study. Study staff will log into a secure system to randomize the participant. The study vaccine associated with that randomization will be selected. A verifier will confirm that the correct vaccine was selected. After verification, study staff will administer the dose.
Masking Description: This is an unblinded, post-licensure study; study staff will not be blinded to participant intervention status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vaxelis (Active Comparator): 165 infants will be randomized to the Vaxelis group, which is licensed for primary vaccination at 2, 4 and 6 months of age.
  Interventions: Drug: Vaxelis
- PedvaxHIB arm (Active Comparator): 165 infants will be randomized to the PedvaxHIB group, which is licensed for primary vaccination at 2 and 4 months of age.
  Interventions: Drug: PedvaxHIB

INTERVENTIONS:
Drug: Vaxelis — Eligible infants will be block randomized to one of two study arms.
  Other Names: Intervention
  Arms: Vaxelis
Drug: PedvaxHIB — Eligible infants will be block randomized to one of two study arms.
  Other Names: Comparator
  Arms: PedvaxHIB arm

SUMMARY:
The main goal of this study is to compare the Haemophilus influenzae type b antibody response in American Indian / Alaska Native (AI/AN) infants to two licensed vaccines: Vaxelis and PedvaxHIB.

DETAILED DESCRIPTION:
Historically, American Indian and Alaska Native (AI/AN) children aged <5 years have experienced invasive H. influenzae type b (Hib) disease at a rate that is at least 5 times higher than the general U.S. population. In the pre-vaccine era, the incidence of Hib disease peaked earlier for AI/AN children at 4-5 months than general US children at 6-9 months. Therefore, prevention efforts for AI/AN populations focused on identifying a vaccine that would protect against disease in early infancy. Studies in AI/AN children revealed that the Hib conjugate vaccine with the capsular polysaccharide (polyribosylribitol phosphate polysaccharide [PRP]) coupled to the outer membrane protein complex of Neisseria meningitidis (OMP) induced anti-PRP IgG titers that correlated with protection (GMC ≥0.15 μg/mL) and demonstrated high efficacy after a single dose in infancy. Hib PRP-OMP was licensed in 1991 as PedvaxHIB; following introduction of a two-dose primary series and a booster dose, the rate of Hib disease decreased substantially among AI/AN children. The importance of PRP-OMP vaccine to disease control was highlighted in the 1990s in Alaska when use of a non-PRP OMP Hib vaccine was associated with an increase in disease incidence in AN children. In 1999, the American Academy of Pediatrics Committee for Native American Child Health released its official preference for Hib PRP-OMP for use in AI/AN populations.

In spite of Hib vaccine coverage similar to or greater than the national average, AI/AN populations periodically experience pediatric cases of invasive Hib disease. In contrast to the pre-Hib vaccine era, a majority of these cases occur in fully vaccinated children beyond the first year of life. This epidemiologic shift in the age at which disease occurs may indicate ongoing transmission in the presence of waning immunity following vaccination.

Vaxelis is a licensed hexavalent combination vaccine that contains Hib PRP-OMP and antigens (Hepatitis B surface antigen, Diphtheria Toxoid, Tetanus Toxoid, Acellular Pertussis [DTaP], and Inactivated Polio Virus [IPV]) to protect against diseases caused by 5 other organisms. Vaxelis contains 3.0 µg/mL of PRP-OMP antigen, compared to 7.5 µg/mL in PedvaxHIB. This lower concentration of PRP-OMP has been shown to be less reactogenic and similarly immunogenic to higher doses. Vaxelis is approved for administration as a 3-dose primary series at 2, 4, and 6 months of age. A booster dose with a different licensed Hib vaccine (e.g., PedvaxHIB, ActHib) is required at 12-15 months. Vaxelis Hib PRP-OMP was found to be highly immunogenic post-dose 2 at 4 months and post-dose 3 at 6 months. However, immunogenicity post-dose 1 was not measured in the phase 3 clinical trials of this vaccine.

In June 2019, the CDC's Advisory Committee on Immunization Practices (ACIP) passed a resolution supporting inclusion of Vaxelis in the Vaccines For Children Program for the general U.S. population. This vaccine was made available for routine use in the U.S. in 2021. A preferential recommendation for use of this vaccine in AI/AN children was not given because post-dose 1 immunogenicity data were not available. To support policy recommendations to protect the health of the AI/AN community, a study is needed to assess non-inferiority of the post-dose 1 immune response to Vaxelis compared to the current recommended product (PedvaxHIB). It is important to demonstrate that infants vaccinated with Vaxelis will be protected early in life, given the historic early peak of Hib disease and the evidence that Hib still circulates in village-based and reservation-based AI/AN communities.

If this study finds that Vaxelis and PedvaxHIB provide comparable protection after one dose, this would support the ACIP making a preferential recommendation for Vaxelis for AI/AN infants. This would expand the options of preferred vaccines for AI/AN infants and potentially provide more long-lasting protection given that 3 doses would be given as part of the primary series.

This study is a prospective, randomized, unblinded, phase IV study of the immunogenicity of two licensed Hib vaccines among AI/AN infants. The study will enroll approximately 330 AI/AN infants on Navajo Nation, on White Mountain Apache (WMA) Tribal lands, and in Anchorage, Alaska who are 6-12 weeks of age and due to receive their first set of routine infant immunizations. Eligible infants whose parents provide written informed consent will be block randomized to one of two study arms - either Vaxelis or PedvaxHIB. Participants will make 5 study visits over the course of approximately 5 months. Participants randomized to the Vaxelis group will receive the vaccination at 2, 4 and 6 months of age, and randomized to the PedvaxHIB group will receive the vaccination at 2 and 4 months of age.

Four blood samples will be collected: at ages 2, 3, 6, and 7 months. These specimens will be tested by ELISA to assess anti-PRP antibody levels. Among infants vaccinated at 2 months of age, the anti-PRP IgG GMC 30 days post dose 1 of Vaxelis will be considered non-inferior if the ratio of the GMC in the Vaxelis group relative to the PedvaxHIB group is >0.67. The statistical criterion we are using to define non-inferiority corresponds to the lower bound of the two-sided 95% confidence interval (CI) on the anti-PRP IgG GMC ratio [Vaxelis / PedvaxHIB] being >0.67. A sample size of 150 evaluable children per group will provide at least 80% power to detect non-inferiority using constrained longitudinal analysis.

Each participant will also be given other routine pediatric immunizations that are not part of the study regimen, per ACIP schedule and recommendations, (e.g., DTaP and IPV at 2, 4 and 6 months, and hepatitis B vaccine at 2 and 6 months, for participants randomized to PedvaxHIB; Prevnar13 at 2, 4 and 6 months, and the rotavirus vaccine series at either 2, 4 and 6 months (if given RotaTeq) or 2 and 4 months (if given Rotarix). Inactivated influenza vaccine will be offered at 6 months of age, as appropriate based on season.

ELIGIBILITY:
Inclusion Criteria:

* Born at gestational age of ≥35 weeks
* AI/AN infant between 6 to 12 weeks of age (42-90 days) at the time of the first vaccination (i.e., Study Day 1)
* Written informed consent provided by parent(s)/Legally Authorized Representative(s) (LARs)
* Investigators believe that the parent(s)/LARs can and will comply with the requirements of the protocol (i.e., return for follow-up visits, recall of adverse events)
* Infant is available to complete the follow-up period of 5 months
* Healthy infant, as established by medical history and clinical examination before entering the study

Exclusion Criteria:

* History of receipt of blood, blood products, or immunoglobulin products since birth or expected receipt through the duration of the study
* Chronic seizure or evolving or unstable neurologic disorder
* Congenital Heart Disease, except for uncomplicated CHD (e.g., PDA, small septal defect)
* Infant of mother with HIV infection
* History of reaction or hypersensitivity likely to be exacerbated by any vaccine component, or to latex
* Infant with confirmed or suspected immunocompromising medical condition, based on medical history, including chronic administration (more than 14 days in the lifetime) of immunosuppressants or other immune-modifying drugs since birth
* Administration of infant vaccines other than birth dose Hepatitis B, prior to the time of enrollment
* Any condition which might interfere with the evaluation of the investigational product, or interpretation of subject safety or study results, in the opinion of the investigator
* Child of an employee of the sponsor, clinical study site, or any other individual involved with the conduct of the study, or an immediate family member of such individuals
* Acute illness and/or fever (temperature ≥100.4 F or ≥38.0 C) at time of enrollment (Note: Participant with fever may be enrolled at later date if symptoms have resolved and all other criteria for inclusion are met at that time)
* Current (or within the past 7 days) or expected receipt of immunosuppressive agents, including steroids, except topical or inhaled steroids (Note: For oral corticosteroids, this will mean prednisone (≥ 0.5 mg/kg/day, or equivalent; participant may be enrolled at a later date if medication use ends and all other criteria for inclusion are met at that time)

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hammitt, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (5):
- United States (5):
  - Alaska Native Medical Center, Anchorage, Alaska
  - Chinle Center for Indigenous Health, Chinle, Arizona
  - Fort Defiance Center for Indigenous Health, Fort Defiance, Arizona
  - Gallup Center for Indigenous Health, Gallup, New Mexico
  - Shiprock Center for Indigenous Health, Shiprock, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vesikari T, Becker T, Vertruyen AF, Poschet K, Flores SA, Pagnoni MF, Xu J, Liu GF, Stek JE, Boisnard F, Thomas S, Ziani E, Lee AW. A Phase III Randomized, Double-blind, Clinical Trial of an Investigational Hexavalent Vaccine Given at Two, Three, Four and Twelve Months. Pediatr Infect Dis J. 2017 Feb;36(2):209-215. doi: 10.1097/INF.0000000000001406. PMID 27846055
- [Background] Bulkow LR, Wainwright RB, Letson GW, Chang SJ, Ward JI. Comparative immunogenicity of four Haemophilus influenzae type b conjugate vaccines in Alaska Native infants. Pediatr Infect Dis J. 1993 Jun;12(6):484-92. doi: 10.1097/00006454-199306000-00006. PMID 8345981
- [Background] Santosham M, Wolff M, Reid R, Hohenboken M, Bateman M, Goepp J, Cortese M, Sack D, Hill J, Newcomer W, et al. The efficacy in Navajo infants of a conjugate vaccine consisting of Haemophilus influenzae type b polysaccharide and Neisseria meningitidis outer-membrane protein complex. N Engl J Med. 1991 Jun 20;324(25):1767-72. doi: 10.1056/NEJM199106203242503. PMID 1903846
- [Background] Singleton R, Bulkow LR, Levine OS, Butler JC, Hennessy TW, Parkinson A. Experience with the prevention of invasive Haemophilus influenzae type b disease by vaccination in Alaska: the impact of persistent oropharyngeal carriage. J Pediatr. 2000 Sep;137(3):313-20. doi: 10.1067/mpd.2000.107843. PMID 10969253
- [Background] Diaz-Mitoma F, Halperin SA, Tapiero B, Hoffenbach A, Zappacosta PS, Radley D, Bradshaw S, Martin JC, Boslego JW, Hesley TM, Bhuyan PK, Silber JL. Safety and immunogenicity of three different formulations of a liquid hexavalent diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine at 2, 4, 6 and 12-14 months of age. Vaccine. 2011 Feb 1;29(6):1324-31. doi: 10.1016/j.vaccine.2010.11.053. Epub 2010 Dec 4. PMID 21134456
- [Background] Silfverdal SA, Icardi G, Vesikari T, Flores SA, Pagnoni MF, Xu J, Liu GF, Stek JE, Boisnard F, Thomas S, Ziani E, Lee AW. A Phase III randomized, double-blind, clinical trial of an investigational hexavalent vaccine given at 2, 4, and 11-12 months. Vaccine. 2016 Jul 19;34(33):3810-6. doi: 10.1016/j.vaccine.2016.05.054. Epub 2016 Jun 18. PMID 27288217
- [Background] State of Alaska Epidemiology Bulletin; Aug 11, 2009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: American Indian and Alaska Native (AI/AN) infants receiving primary care at five Indian Health Service (IHS)/Tribal Health facilities in Alaska and the Navajo Nation were recruited from December 2021 to April 2023. The first participant was enrolled in January 2022.
Pre-assignment Details: 1736 infants were screened for eligibility and 333 infants were enrolled in the study.
Groups:
- PedvaxHIB Arm: 166 infants will be randomized to the PedvaxHIB group, which is licensed for primary vaccination at 2 and 4 months of age.
  PedvaxHIB: Eligible infants will be block randomized to one of two study arms.
- Vaxelis: 167 infants will be randomized to the Vaxelis group, which is licensed for primary vaccination at 2, 4 and 6 months of age.
  Vaxelis: Eligible infants will be block randomized to one of two study arms.
Period: Overall Study
Arm/Group | PedvaxHIB Arm | Vaxelis
Started | 166 | 167
Completed | 144 | 152
Not Completed | 22 | 15

BASELINE CHARACTERISTICS:
Groups:
- PedvaxHIB Arm: Participants received 0.5 mL doses of PedvaxHIB® (7.5 µg/mL PRP-OMP) administered intramuscularly at age 2 months and 4 months along with their other routine immunizations according to the U.S. vaccination schedule for children.
- Vaxelis: Participants received 0.5 mL doses of Vaxelis® (3.0 µg/mL PRP-OMP + diphtheria, tetanus, pertussis [acellular, component], poliomyelitis [inactivated], and hepatitis B [recombinant deoxyribonucleic acid (rDNA)) administered intramuscularly at age 2 months, 4 months and 6 months along with their other routine immunizations according to the U.S. vaccination schedule for children.
- Total: Total of all reporting groups
Arm/Group | PedvaxHIB Arm | Vaxelis | Total
Number analyzed (Participants) | 166 | 167 | 333
Age, Continuous [Median (Inter-Quartile Range); unit: Days] | 59 [45 to 63] | 60 [46 to 63] | 60 [46 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 83 | 175
  Male | 74 | 84 | 158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 166 | 167 | 333
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Anti-PRP IgG Geometric Mean Concentration (GMC)
Description: The non-inferiority of the anti-PRP IgG Geometric Mean Concentration (GMC) 30 days after dose 1 of Vaxelis administered at 2 months of age, compared to PedvaxHIB. GMC was modeled using constrained longitudinal analysis (cLDA) of anti-PRP IgG concentration at all study visits.
Time Frame: 30 days after dose 1
Population: All specimens were included for which valid concentration results were obtained adhering to study procedures and intervals between primary doses, as defined in the protocol. Participants with incomplete data for the time series contribute their available data to the overall model.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | PedvaxHIB Arm | Vaxelis
Number analyzed (Participants) | 163 | 167
μg/mL | 0.40 [0.31 to 0.5] | 0.41 [0.33 to 0.51]
Statistical Analysis 1: Comparison: PedvaxHIB Arm vs Vaxelis; Test type: Non-Inferiority — The anti-PRP IgG GMC for children receiving dose 1 of Vaxelis® was defined a priori as non-inferior if it was within a 1.5-fold margin of the GMC for children receiving dose 1 of PedvaxHIB®, corresponding to the lower bound of the 95% confidence interval (CI) of the IgG GMC ratio (Vaxelis® to PedvaxHIB®) being greater than 0.67; p = 0.85, Constrained Longitudinal Analysis; Ratio of Geometric Mean Concentration = 1.03, 95% CI 2-sided [0.75 to 1.41] — The lower bound of the 95% confidence interval was greater than the pre-specified non-inferiority margin of 0.67. Thus, Vaxelis® post-dose 1 anti-PRP IgG immunogenicity met the non-inferiority criterion compared to PedvaxHIB®

2. Secondary Outcome: Percent of Anti-PRP IgG ≥0.15 µg/mL 30 Days After Dose 1
Description: Describe the percent of infants with anti-PRP IgG ≥0.15 µg/mL 30 days after dose 1 of Vaxelis or PedvaxHIB.
Time Frame: 30 days after dose 1 of Vaxelis or PedvaxHIB
Population: All specimens from which valid concentration measurements were made from participants adhering to study procedures and intervals between primary doses, as defined in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | PedvaxHIB Arm | Vaxelis
Number analyzed (Participants) | 146 | 152
Participants | 104 | 115
Statistical Analysis 1: Comparison: PedvaxHIB Arm vs Vaxelis; Test type: Other; p = 0.39, Chi-squared

3. Secondary Outcome: Percent of Anti-PRP IgG ≥1.0 µg/mL 30 Days After Dose 1
Description: Describe the percent of infants with anti-PRP IgG ≥1.0 µg/mL 30 days after dose 1 of Vaxelis or PedvaxHIB.
Time Frame: 30 days after dose 1 of Vaxelis or PedvaxHIB
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PedvaxHIB Arm | Vaxelis
Number analyzed (Participants) | 146 | 152
Participants | 40 | 38
Statistical Analysis 1: Comparison: PedvaxHIB Arm vs Vaxelis; Test type: Other; p = 0.64, Chi-squared

4. Secondary Outcome: Percent of Anti-PRP IgG ≥0.15 µg/mL on Day 121
Description: Describe the percent of infants with anti-PRP IgG ≥0.15 µg/mL on Day 121 after initiation of the primary series, i.e., 60 days after dose 2 of Vaxelis and dose 2 of PedvaxHIB.
Time Frame: 60 days after dose 2 of Vaxelis and dose 2 of PedvaxHIB
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PedvaxHIB Arm | Vaxelis
Number analyzed (Participants) | 122 | 133
Participants | 115 | 126
Statistical Analysis 1: Comparison: PedvaxHIB Arm vs Vaxelis; Test type: Other; p = 0.87, Chi-squared

5. Secondary Outcome: Percent of Anti-PRP IgG ≥1.0 µg/mL on Day 121
Description: Describe the percent of infants with anti-PRP IgG ≥1.0 µg/mL on Day 121 after initiation of the primary series, i.e., 60 days after dose 2 of Vaxelis and dose 2 of PedvaxHIB.
Time Frame: 60 days after dose 2 of Vaxelis and dose 2 of PedvaxHIB
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PedvaxHIB Arm | Vaxelis
Number analyzed (Participants) | 122 | 133
Participants | 100 | 102
Statistical Analysis 1: Comparison: PedvaxHIB Arm vs Vaxelis; Test type: Other; p = 0.3, Chi-squared

6. Secondary Outcome: Percent of Anti-PRP IgG ≥0.15 µg/mL on Day 151
Description: Describe the percent of infants with anti-PRP IgG ≥0.15 µg/mL on Day 151 after initiation of the primary series, i.e., 30 days after dose 3 of Vaxelis and 90 days after dose 2 of PedvaxHIB.
Time Frame: 30 days after dose 3 of Vaxelis and 90 days after dose 2 of PedvaxHIB
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PedvaxHIB Arm | Vaxelis
Number analyzed (Participants) | 117 | 128
Participants | 106 | 122
Statistical Analysis 1: Comparison: PedvaxHIB Arm vs Vaxelis; Test type: Other; p = 0.15, Chi-squared

7. Secondary Outcome: Percent of Anti-PRP IgG ≥1.0 µg/mL on Day 151
Description: Describe the percent of infants with anti-PRP IgG ≥1.0 µg/mL on Day 151 after initiation of the primary series, i.e., 30 days after dose 3 of Vaxelis and 90 days after dose 2 of PedvaxHIB.
Time Frame: 30 days after dose 3 of Vaxelis and 90 days after dose 2 of PedvaxHIB
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PedvaxHIB Arm | Vaxelis
Number analyzed (Participants) | 117 | 128
Participants | 84 | 107
Statistical Analysis 1: Comparison: PedvaxHIB Arm vs Vaxelis; Test type: Other; p = 0.03, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 7 months post first dose of study vaccine
Description: SAEs were assessed via parental questionnaire and chart review at each study visit. SAEs were assessed for severity and causality by the Investigators. Non-serious adverse events were not monitored.
Arm/Group | PedvaxHIB Arm | Vaxelis
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/167
Serious Adverse Events (participants affected / at risk) | 12/166 | 9/167
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PedvaxHIB Arm (N=166) | Vaxelis (N=167)
Acute gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Broken Femur (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 4 (4)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Serizure, or seizure-like activity (Nervous system disorders) | 0 (0) | 2 (2)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Viral illness with hypoxia (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT04978818/Prot_SAP_000.pdf